CLINICAL TRIAL: NCT00836823
Title: The Long Term Effects of Alfuzosin (Xatral XL) in LUTS/BPH Patients: Evaluation of Symptom-specific Goal Achievement According to Symptom Improvement, Bladder Outlet Obstruction Grade and Bladder Contractility
Brief Title: Evaluation of Symptom-specific Goal Achievement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-10-044
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: Patient-reported most bothersome symptom; Patient-reported symptom-specific goal achievement; Medical treatment
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Alpha blocker (Experimental): Alfuzosin 10mg
  Interventions: Drug: Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin — Alfuzosin 10mg once daily for 12 months
  Other Names: XATRAL XL

SUMMARY:
Lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH) consists of a constellation of symptoms (including voiding, storage, and post-micturition). The impact of the LUTS on patients' health-related quality of life is substantial and multifaceted. Thus, the therapies aimed at treating BPH are concerned primarily with improving patients' symptoms, thereby improving quality of life. When multiple symptoms are present, the level of bother associated with individual symptoms varies and patients prioritize their treatment goals for symptom relief. A measure that addresses patients' most bothersome symptoms (MBS) and evaluation of symptom-specific goal achievements may lead to improved outcomes and patient satisfaction to the treatment. The objectives of this study were (1) to assess patient-reported MBS and symptom-specific goal achievements (PGA) with medical treatment in BPH patients, and (2) to identify factors that influence or have relation to the PGA.

ELIGIBILITY:
Inclusion Criteria:

* males ≥50 years with LUTS secondary to BPH
* Moderate to severe LUTS : IPSS ≥ 8
* An enlarged prostate : TRUS ≥25 mL
* Decreased peak flow rate : Qmax ≤15mL/s (volume voided ≥ 120 mL)
* Having signed the informed consent to participate in the study.

Exclusion Criteria:

* Post voided residual urine ≥ 200mL
* Patients performing catheterization
* Urinary tract infection patients
* Patients taking 5 alpha reductase inhibitor
* Known hypersensitivity to alfuzosin
* History of postural hypotension or syncope
* Hypertension patients treated with other alpha1-blockers
* Patients newly taking anticholinergic medication within 1 month
* Hepatic insufficiency (AST/ALT ≥ 2 times of normal range)
* Renal insufficiency (s-Cr ≥ 2mg/dL)
* Unstable angina pectoris
* Uninvestigated hematuria
* Serum PSA ≥ 4 ng/mL (biopsy proven no cancer patients can be included)
* Interstitial cystitis patients
* Severe concomitant condition threatening life.
* Patient who is unable to make voiding diary
* Bladder or prostate cancer patients
* Patients receiving prostate or bladder surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Patient-reported goal achievements for the most bothersome symptoms | 12 months of treatment

SECONDARY OUTCOMES:
Patient-reported goal achievement for the most bothersome symptom using Likert scale | 3, 6, and 12 months of treatment
Changes in: IPSS, ICS-male questionnaire, maximal flow rate, post-voided residual urine, voiding chart parameters | 3, 6, and 12 months of treatment
Global impression of improvement | 3, 6, and 12 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (2):
- South Korea (2):
  - Asan Medical Center, Ulsan College of Medicine, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Lee YS, Lee HN, Han JY, Choo MS, Lee KS. Most bothersome symptom and symptom specific goal achievement in patients with benign prostatic obstruction: a prospective open label study. J Urol. 2011 Mar;185(3):1003-9. doi: 10.1016/j.juro.2010.10.085. Epub 2011 Jan 19. PMID 21251673